CLINICAL TRIAL: NCT02245854
Title: Efficacy and Safety of a New Polypectomy Snare for Cold-polypectomy for Subcentimetric Colorectal Polyps: the E-scope (Efficacy and Safety of COld PolypEctomy) Trial
Brief Title: Efficacy and Safety of a New Polypectomy Snare for Cold-polypectomy for Small Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: San Gerardo Hospital (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Responsible of the Clinical Research Project, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-Scope
Record Dates: First submitted 2014-09-01; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Polyp of Large Intestine; Colonic Polyps; Colon Nos Polypectomy Tubular Adenoma; Complications; Bleeding
Keywords: diminutive polyps; small polyps; cold snare polypectomy; complications; bleeding
MeSH Terms: conditions — Colonic Polyps; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colonic polyps (Experimental): Exacto™
  Interventions: Device: Exacto™

INTERVENTIONS:
Device: Exacto™ — Cold snare polypectomy

SUMMARY:
Colorectal cancer is a major cause of morbidity and mortality in Western countries. Scientific studies have shown that endoscopic polypectomy is efficacious in preventing CRC incidence and mortality.

Endoscopic polypectomy carries a risk of major complications, such as bleeding or bowel perforation, so that a careful balance between efficacy and safety appears to be clinically relevant.

Most of the polypectomies are performed for diminutive (<5 mm) or small (6-9 mm) lesions, which represent over 90% of all the polyps.

To minimize the risk of complications when removing <10 mm polyps, cold-polypectomy techniques - i.e. without electric current - by means of biopsy forceps or snare, have been proposed.

Although the risk of perforation is virtually excluded by cold-polypectomy, the lack of electrocautery may result in an increased risk of bleeding. The safety of cold-snare polypectomy has however been recently shown in controlled trials.

Regarding the efficacy of cold-polypectomy for subcentimetric polyps, very few studies have assessed the post-polypectomy completeness of the removal of polyp tissue (i.e. residual disease), and no studies have compared it to conventional polypectomy.

The investigators perform this study to assess both the efficacy and safety of a novel snare (Exacto™) for polyp removal.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing colonoscopy, with at least one and no more than 5 polyps <10 mm.
* The patient is at satisfactory risk to undergo abdominal surgery.
* The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

* Patients with inflammatory bowel disease.
* Patients undergoing standard snare resection (with cautery) of polyps larger than 10 mm.
* Patients with a personal history of polyposis syndrome.
* Patients with suspected chronic stricture potentially precluding complete colonoscopy.
* Patients with diverticulitis or toxic megacolon.
* Patients with a history of radiation therapy to abdomen or pelvis.
* Patients with a history of severe cardiovascular, pulmonary, liver or renal disease.
* Personal history of coagulation disorders or use of anticoagulants/clopidogrel/aspirin/ticlopidine.
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of complete polyp removal | One year
  Clinical success, defined as absence of polyp tissue, either hyperplastic or adenomatous, on the margins of the polypectomy area after cold-polypectomy of subcentimetric polyps. Such assessment is performed on two biopsies performed on the polypectomy scar. The investigators will calculate the percentage (%) of complete and incomplete polypectomies with the new device.

SECONDARY OUTCOMES:
Clinical success according to size | One year
  Clinical success (as defined in the primary end-point) according to the size class: diminutive (<5 mm) and small (6-9 mm) polyps.
Post-polypectomy bleeding rates | One year
  Post-polypectomy bleeding defined as any bleeding requiring immediate therapeutic endoscopic procedure (i.e. clipping, electrocautery) or delayed treatment, such as hospitalization or new endoscopic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (3):
- Italy (3):
  - Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milan, Italy
  - San Gerardo Hospital, Monza
  - Azienda Ospedaliera "Maggiore della Carità", Novara

REFERENCES:
- [Background] Repici A, Hassan C, Vitetta E, Ferrara E, Manes G, Gullotti G, Princiotta A, Dulbecco P, Gaffuri N, Bettoni E, Pagano N, Rando G, Strangio G, Carlino A, Romeo F, de Paula Pessoa Ferreira D, Zullo A, Ridola L, Malesci A. Safety of cold polypectomy for <10mm polyps at colonoscopy: a prospective multicenter study. Endoscopy. 2012 Jan;44(1):27-31. doi: 10.1055/s-0031-1291387. Epub 2011 Nov 28. PMID 22125197
- [Background] Ichise Y, Horiuchi A, Nakayama Y, Tanaka N. Prospective randomized comparison of cold snare polypectomy and conventional polypectomy for small colorectal polyps. Digestion. 2011;84(1):78-81. doi: 10.1159/000323959. Epub 2011 Apr 14. PMID 21494037
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514
- [Background] Paspatis GA, Tribonias G, Konstantinidis K, Theodoropoulou A, Vardas E, Voudoukis E, Manolaraki MM, Chainaki I, Chlouverakis G. A prospective randomized comparison of cold vs hot snare polypectomy in the occurrence of postpolypectomy bleeding in small colonic polyps. Colorectal Dis. 2011 Oct;13(10):e345-8. doi: 10.1111/j.1463-1318.2011.02696.x. PMID 21689363
- [Background] Lieberman D, Moravec M, Holub J, Michaels L, Eisen G. Polyp size and advanced histology in patients undergoing colonoscopy screening: implications for CT colonography. Gastroenterology. 2008 Oct;135(4):1100-5. doi: 10.1053/j.gastro.2008.06.083. Epub 2008 Jul 3. PMID 18691580
- [Background] Heldwein W, Dollhopf M, Rosch T, Meining A, Schmidtsdorff G, Hasford J, Hermanek P, Burlefinger R, Birkner B, Schmitt W; Munich Gastroenterology Group. The Munich Polypectomy Study (MUPS): prospective analysis of complications and risk factors in 4000 colonic snare polypectomies. Endoscopy. 2005 Nov;37(11):1116-22. doi: 10.1055/s-2005-870512. PMID 16281142
- [Background] Panteris V, Haringsma J, Kuipers EJ. Colonoscopy perforation rate, mechanisms and outcome: from diagnostic to therapeutic colonoscopy. Endoscopy. 2009 Nov;41(11):941-51. doi: 10.1055/s-0029-1215179. Epub 2009 Oct 28. PMID 19866393
- [Background] Atkin WS, Edwards R, Kralj-Hans I, Wooldrage K, Hart AR, Northover JM, Parkin DM, Wardle J, Duffy SW, Cuzick J; UK Flexible Sigmoidoscopy Trial Investigators. Once-only flexible sigmoidoscopy screening in prevention of colorectal cancer: a multicentre randomised controlled trial. Lancet. 2010 May 8;375(9726):1624-33. doi: 10.1016/S0140-6736(10)60551-X. Epub 2010 Apr 27. PMID 20430429